CLINICAL TRIAL: NCT03803228
Title: Comparison of the Cumulative Number of Oocytes Obtained With 2 Controlled Ovarian Hyperstimulations (COH) Within the Same Cycle With FertistartKit® (DUOSTIM) Versus 2 Conventional COH in Poor Ovarian Responders Undergoing IVF. Bistim Study
Brief Title: Dual Ovarian Stimulation (DUOSTIM) for Poor Ovarian Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Laboratoires Genévrier (Industry); IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BISTIM
Record Dates: First submitted 2018-08-08; First posted 2019-01-14 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DUOSTIM (Experimental): (stim 1) flexible antagonist protocol with pre-treatment with estrogen (S1 between J1 and J8 under E2) and stimulation with Fertistartkit® 300 IU / d; triggering by rHCG (Ovitrelle®250μg) and puncture at 36h; oocyte freezing; (stim 2) resumption of stimulation only by Fertistratkit® 300 IU / day from the day after the puncture; introduction of Progestan® 7 days later to avoid menstruation during the second puncture; triggering with rHCG and second puncture at 36h associated with the devitrification of stim 1 oocytes, with sperm collection and embryonic vitrification. Transfer of frozen embryos to the subsequent cycle in the natural cycle (without HCG) and until the frozen embryos are exhausted.
  Interventions: Drug: DUOSTIM
- Conventional stimuli (Active Comparator): (stim 1) flexible antagonist protocol with pre-treatment with estrogen (S1 between J1 and J8 under E2) and stimulation with Fertistartkit® 300 IU / d; triggering by rHCG (Ovitrelle®250μg) and puncture at 36h; fresh embryonic transfer if satisfactory endometrial conditions with luteal phase support by vaginal micronized progesterone Progestan® 600 mg / d; otherwise embryonic freezing and transfer of frozen embryos to the subsequent cycle in the natural cycle until the frozen embryos are exhausted.
  (stim 2) ditto starting on the next cycle if possible or the next one. Hormonal Controls + Ultrasound During Stimulation: Blocking / S1 - S5 / S6 - S8 / S9 - SHCG / SHCG-1
  Interventions: Drug: Conventional stimuli

INTERVENTIONS:
Drug: DUOSTIM — 2 consecutive stimulations by Fertistartkit® on the same cycle
  Other Names: Same monthly cycle
  Arms: DUOSTIM
Drug: Conventional stimuli — 2 stimulations by Fertistartkit® performed on 2 different cycles
  Other Names: Two different menstrual cycles
  Arms: Conventional stimuli

SUMMARY:
During ovarian stimulation, all the follicles grow under the action of FSH, only the selected follicles and with the faster growth are taken. However during this stimulation, other smaller follicles are also recruited and sensitized, which may increase the selection of follicles available on the follicular wave following. In patients with weak reserve this potentiation has a great interest, and the sequence of 2 stimulations on the same cycle could make it possible to obtain a larger number of oocytes and embryos, thus giving a better chance of delivery than on 2 distinct cycles of stimulation. However, this is preliminary data that needs to be confirmed with a randomized controlled trial. In this population of poor prognosis, the use of FSH-associated LH activity may optimize the ovarian response to stimulation, particularly the combination containing placental HCG (Fertistartkit®) that obtaining a slightly higher number of oocytes than highly purified HMG (Menopur®).

DETAILED DESCRIPTION:
Ovarian stimulation is an essential prerequisite for any in vitro fertilization attempt (IVF) to optimize the chances of delivery per cycle. These depend in the first place on the age of the patients and secondly on the number of oocytes collected. There is a strong correlation between these two factors, the ovarian reserve diminishing with age. In older patients or patients with decreased reserve, however, the number of oocytes collected remains a prognostic factor for the chances of delivery.

At the present time, there is no validated intervention that would bring a significant interest on the number of oocytes obtained in the group of bad responder patients. However, it is a very heterogeneous population whose definition has been proposed only recently, the Bologna criteria and questioned by a new proposal from the Poseidon group. The latter is more focused on the prognosis of success, differentiating patients with a diminished reserve (count of antral follicles CFA <5 and / or AMH <1.2 ng / ml) from those with an "unexpected" bad response. As the profiles are better defined, it is easier to determine the impact of a strategy in a specific group.

Recent clarifications on the ovarian cycle and folliculogenesis have shown that several waves of follicular development coexist on the same cycle and that it is perfectly possible to obtain a follicular development with a luteal phase equivalent oocyte quality, compared to conventional stimulations performed in the follicular phase. The main constraint of luteal phase stimulation is the lack of possibility of fresh transfer due to non-synchronization with the endometrium. This constraint is today secondary given the evolution of conservation techniques with the development of embryonic and oocyte vitrification.

On the other hand, there is a differential dependence of FSH follicles, their sensitivity depending on the number of FSH receptors and their duration of exposure to FSH. During ovarian stimulation, all the follicles grow under the action of FSH, only the selected follicles and with the faster growth are taken. However during this stimulation, other smaller follicles are also recruited and sensitized, which may increase the selection of follicles available on the follicular wave following. In patients with weak reserve this potentiation has a great interest, and the sequence of 2 stimulations on the same cycle could make it possible to obtain a larger number of oocytes and embryos, thus giving a better chance of delivery than on 2 distinct cycles of stimulation. However, this is preliminary data that needs to be confirmed with a randomized controlled trial. In this population of poor prognosis, the use of FSH-associated LH activity may optimize the ovarian response to stimulation, particularly the combination containing placental HCG (Fertistartkit®) that obtaining a slightly higher number of oocytes than highly purified HMG (Menopur®).

ELIGIBILITY:
Inclusion Criteria:

* Women from 20 to 41 years old
* CFA <5 and / or AMH <1, 2 ng / ml
* 19 ≤ BMI ≤ 32
* Supports IVF or ICSI
* If antecedent IVF / ICSI, number of oocytes collected <4
* Attack rank (puncture with transfer) <3
* Affiliation to the general social security scheme and benefiting from 100% infertility

Exclusion Criteria:

* Confirmed ovarian insufficiency (amenorrhea)
* FSH> 20 IU / l or CFA <1
* Puncture rank> 3
* Azoospermia or cryptozoospermia
* Against indication to ovarian stimulation
* Presence of a cyst of indeterminate etiology, ovarian, uterine or mammary carcinoma, hypothalamic or pituitary tumors
* Hypersensitivity to any of the medicines in the protocol
* Moderate or severe pathology of renal or hepatic function
* Evolutionary thromboembolic accidents

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
cumulative number of oocytes on 2 punctures | up to 60 days
  cumulative number of oocytes on 2 punctures

SECONDARY OUTCOMES:
cumulative number of follicles> 14mm | up to 60 days
  cumulative number of follicles> 14mm
cumulative number of oocytes in metaphase II | up to 60 days
  cumulative number of oocytes in metaphase II
cumulative number of embryos obtained | 1 month
  cumulative number of embryos obtained
number of embryos transferred | up to 60 days
  number of embryos transferred
number of frozen embryos | 1.5 month
  number of frozen embryos
dose of FSH | up to 60 days
  cumulative total dose of FSH
the number of stimulation days | up to 20 days
  the number of stimulation days
estradiol level | up to 20 days
  estradiol level
LH level | up to 20 days
  LH level
progesterone level | up to 20 days
  progesterone level
transfer rate | 3 months
  cancellation or no transfer rate
rates of early pregnancy | up to 9 months
  cumulative rates of early pregnancy (HCG> 100) and ultrasound (6-7SA)
number of beginner pregnancy | up to 9 months
  number of beginner pregnancy in each groups
cumulative cost | up to 9 months
  cumulative cost of 2 attempts including frozen embryo transfers (treatments, consultations, MPA laboratory and monitoring exams)
Side effects | up to 9 months
  reported side effects

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie MASSIN, MD, Principal Investigator — CHI Créteil
Locations (4):
- France (4):
  - Polyclinique Jean Villar, Bruges
  - CHI Creteil, Créteil
  - Cabinet Médical Carré Saint Giniez, Marseille
  - Polyclinique Saint Roch, Montpellier

REFERENCES:
- [Derived] Massin N, Abdennebi I, Porcu-Buisson G, Chevalier N, Descat E, Pietin-Vialle C, Goro S, Brussieux M, Pinto M, Pasquier M, Bry-Gauillard H. The BISTIM study: a randomized controlled trial comparing dual ovarian stimulation (duostim) with two conventional ovarian stimulations in poor ovarian responders undergoing IVF. Hum Reprod. 2023 May 2;38(5):927-937. doi: 10.1093/humrep/dead038. PMID 36864699